## Feasibility and acceptability of six-weeks of high intensity interval training in wheelchair users with SCI

**Short Title:** HIIT in Spinal Cord Injury (HIIT-SCI)

**Principal Investigator:** Alicia Koontz, PhD, RET

Human Engineering Research Laboratories

VA Pittsburgh HealthCare System

University of Pittsburgh 6425 Penn Avenue, Suite 400 Pittsburgh, PA 15206-4022 Phone: 412-822-3700

Funded By: University of Alabama – Birmingham

1720 University Blvd Birmingham, AL 35294

(205) 934-4011

Eunice Kennedy Shriver National Institute of Child Health and

Human Development (NICHD)

NIH Clinical Center

10 Center Dr

Bethesda, MD 20814

**Study Protocol Number**: NCT03152110 (National Clinical Trials)

PRO17020277 (OSIRIS)

STUDY19040142 (University of Pittsburgh)

IRB last modified: 16 April 2020

## Statistical Analysis Plan

Distributions of all data will be examined. Should outliers or distributions that are nonlinear in nature be present, appropriate transformations will be performed. Means and standard deviations, or medians and ranges, as appropriate, will be calculated for all variables. Total number of training sessions completed and numbers of sessions meeting criteria for HIIT target intensity (e.g. average power achieved over work phases) will be determined to evaluate feasibility. A paired t-test will be used to compare the primary outcome measures obtained during the pre and post exercise max testing (i.e. physical capacity measures [peak power, peak VO<sub>2</sub><sup>+</sup>, time to exhaustion].

IRB last modified: 16 April 2020